CLINICAL TRIAL: NCT00090402
Title: Fish Oil and Alpha Lipoic Acid in Mild Alzheimer's Disease
Brief Title: Fish Oil and Alpha Lipoic Acid in Treating Alzheimer's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Lynne Shinto, ND, MPH, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IA0062; 1R21AG023805-01 (NIH); 5R21AG023805-02 (NIH); AG08017 (Other Grant/Funding Number: National Institute of Aging); M01RR000334 (NIH)
Record Dates: First submitted 2004-08-25; First posted 2004-08-26 (Estimated); Results first posted 2010-02-26 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-06

CONDITIONS: Alzheimer's Disease; Oxidative Stress; Dementia; Hyperlipidemia; Inflammation
Keywords: Fish Oils; Thioctic Acid; Antioxidants; Dietary Supplements
MeSH Terms: conditions — Alzheimer Disease; Dementia; Hyperlipidemias; Inflammation | interventions — Fish Oils; Fatty Acids, Omega-3; Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fish Oil Placebo & Lipoic Acid Placebo (Placebo Comparator): Three 1-gram placebo-fish oil capsules (2 in the morning, 1 evening) plus one 600 milligram placebo-lipoic acid per day. Placebo fish oil capsules consisted of soybean oil flavored with lemon flavor and 5% fish oil to match fish oil capsules. LA placebo contained no LA and the following excipients: lactose, hypromellose, silicon dioxide, microcrystalline cellulose, polyethylene glycol, povidone, corn starch, talc, and magnesium stearate.
  Interventions: Other: Fish Oil Placebo; Other: Lipoic Acid Placebo
- Fish Oil Only (Active Comparator): Three 1-gram fish oil concentrate capsules in triglyceride form (675 milligrams DHA and 975 milligrams EPA), 2 in the morning and 1 in the evening, plus one 600 milligram placebo-lipoic acid (containing no LA and the following excipients: lactose, hypromellose, silicon dioxide, microcrystalline cellulose, polyethylene glycol, povidone, corn starch, talc, and magnesium stearate) per day.
  Interventions: Dietary Supplement: Fish Oil; Other: Lipoic Acid Placebo
- Fish Oil Plus Lipoic Acid (Experimental): Three 1-gram placebo-fish oil capsules (2 in the morning, 1 evening) plus one 600 milligram lipoic acid (LA) capsule in the racemic form per day.
  Interventions: Dietary Supplement: Fish Oil; Dietary Supplement: Lipoic Acid

INTERVENTIONS:
Dietary Supplement: Fish Oil — Fish oil capsule
  Other Names: Fish oil concentrate, omega-3 fatty acids
  Arms: Fish Oil Only; Fish Oil Plus Lipoic Acid
Dietary Supplement: Lipoic Acid — Lipoic acid capsule
  Other Names: thiotic acid, alpha lipoic acid
  Arms: Fish Oil Plus Lipoic Acid
Other: Fish Oil Placebo — Soybean oil placebo capsule
  Other Names: Placebo (for fish oil)
  Arms: Fish Oil Placebo & Lipoic Acid Placebo
Other: Lipoic Acid Placebo — Lipoic acid (LA) placebo capsule containing no LA
  Other Names: Placebo (for lipoic acid)
  Arms: Fish Oil Only; Fish Oil Placebo & Lipoic Acid Placebo

SUMMARY:
The purpose of this study is to determine the effect of fish oil and the antioxidant alpha lipoic acid on factors in the blood that are associated with the progression of Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a serious condition associated with increased inflammation, cholesterol, and oxidative stress (a condition involving an excess of free radicals and a decrease in antioxidant levels). Fish oil and alpha lipoic acid, which have few side effects, may help relieve these problems; therefore, these supplements may slow the progression of AD, particularly when given in combination. This study will evaluate the effect of fish oil and alpha lipoic acid on inflammation, lipid levels, and oxidative stress.

Participants in this study will be randomly assigned to receive fish oil alone, fish oil and alpha lipoic acid, or placebo for 1 year. AD rating scales as well as urine and blood tests will be used to assess participants. Participants will have monthly clinic visits during the study to monitor adverse events and to undergo various laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer's Disease or mild cognitive impairment
* Mini Mental State Examination (MMSE) score between 18 and 26
* Clinical Dementia Rating (CDR) of 0.5 or 1.0
* Fluent in English

Exclusion Criteria:

* Use of lipid lowering medications
* Consumption of fish of more than twice a week
* Use of omega and alpha lipoic acid supplements
* Use of systemic corticosteroids, neuroleptics, anti-Parkinsonian agents, or narcotic analgesics
* Depression
* Any other serious health conditions that may interfere with the study
* Enrollment in another clinical trial

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-04 (Actual); Primary Completion 2006-01-03 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynne H. Shinto, ND, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calon F, Lim GP, Yang F, Morihara T, Teter B, Ubeda O, Rostaing P, Triller A, Salem N Jr, Ashe KH, Frautschy SA, Cole GM. Docosahexaenoic acid protects from dendritic pathology in an Alzheimer's disease mouse model. Neuron. 2004 Sep 2;43(5):633-45. doi: 10.1016/j.neuron.2004.08.013. PMID 15339646
- [Background] Morris MC, Evans DA, Bienias JL, Tangney CC, Bennett DA, Wilson RS, Aggarwal N, Schneider J. Consumption of fish and n-3 fatty acids and risk of incident Alzheimer disease. Arch Neurol. 2003 Jul;60(7):940-6. doi: 10.1001/archneur.60.7.940. PMID 12873849
- [Background] Lovell MA, Xie C, Xiong S, Markesbery WR. Protection against amyloid beta peptide and iron/hydrogen peroxide toxicity by alpha lipoic acid. J Alzheimers Dis. 2003 Jun;5(3):229-39. doi: 10.3233/jad-2003-5306. PMID 12897407
- [Result] Shinto L, Quinn J, Montine T, Dodge HH, Woodward W, Baldauf-Wagner S, Waichunas D, Bumgarner L, Bourdette D, Silbert L, Kaye J. A randomized placebo-controlled pilot trial of omega-3 fatty acids and alpha lipoic acid in Alzheimer's disease. J Alzheimers Dis. 2014;38(1):111-20. doi: 10.3233/JAD-130722. PMID 24077434

RESULTS

PARTICIPANT FLOW:
Groups:
- Fish Oil: Fish oil concentrate, daily dose 3 grams per day containing 675 mg docosahexanoic acid and 975 mg eicosapentanoic acid, taken for 12 months.
- Placebo: Placebo oil (soybean oil), daily dose 3 grams taken for 12 months
- Fish Oil Plus Lipoic Acid: Fish oil concentrate, daily dose 3 grams per day containing 675 mg docosahexaenoic acid and 975 mg eicosapentanoic acid plus alpha lipoic acid (racemic) daily dose 600 mg taken for 12 months.
Period: Overall Study
Arm/Group | Fish Oil | Placebo | Fish Oil Plus Lipoic Acid
Started | 13 | 13 | 13
Completed | 11 | 11 | 12
Not Completed | 2 | 2 | 1
Not completed — Death | 1 | 1 | 0
Not completed — subject moved | 0 | 1 | 0
Not completed — stopped taking study medication | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Fish Oil: Fish oil concentrate, daily dose 3 grams per day containing 675 mg docosahexaenoic acid and 975 mg eicosapentanoic acid, taken for 12 months.
- Total: Total of all reporting groups
Arm/Group | Placebo | Fish Oil | Fish Oil Plus Lipoic Acid | Total
Number analyzed (Participants) | 13 | 13 | 13 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3 | 6
  >=65 years | 11 | 12 | 10 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.2 (10.8) | 75.9 (8.1) | 76.7 (10.6) | 75.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 6 | 21
  Male | 6 | 5 | 7 | 18
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 13 | 39

OUTCOME MEASURES:

1. Primary Outcome: F2-isoprostane Level Urine F2-Isoprostanes
Description: F2-isoprostane is a biomarker was used as an effective indicator for detecting a decrease in systemic oxidative damage (oxidative damage in lipids). Urine F2-Isoprostanes were used to avoid ex vivo lipid peroxidation that can occur with plasma samples.
Time Frame: baseline, 12 months
Population: intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: nanogram per miligram
Arm/Group | Placebo | Fish Oil | Fish Oil Plus Lipoic Acid
Number analyzed (Participants) | 13 | 13 | 13
nanogram per miligram | 0.40 (1.10) | -2.02 (3.30) | 0.45 (0.53)
Statistical Analysis 1: Comparison: Placebo vs Fish Oil vs Fish Oil Plus Lipoic Acid; Test type: Superiority or Other; p = 0.83, Regression, Linear; Adjusted for age and body mass index

2. Primary Outcome: Change in Mini-Mental State Exam (MMSE) Score From Baseline to 12 Months
Description: The MMSE is a measure of global cognitive function, and scores range from 0-30, with a lower score indicates greater cognitive impairment.
Time Frame: baseline, 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Fish Oil | Fish Oil Plus Lipoic Acid
Number analyzed (Participants) | 11 | 11 | 12
units on a scale | -4.64 (4.65) | -4.27 (4.15) | -1.00 (2.30)

3. Secondary Outcome: Change in Activities of Daily Living/Instrumental Activities of Daily Living (ADL/IADL) Scores From Baseline to 12 Months
Description: The Activities of Daily Living/Instrumental Activities of Daily Living (ADL/IADL) measures an individual's ability to carry out tasks that are important for daily living and capture functional changes. Scores for each question range from 0 (no assistance needed) to 2 (full assistance needed), and were assessed by informant interview. The combination of scores for ADL (ranging from 0-18) and IADL (0-14) is the outcome (0-32), with higher scores indicating lesser ability to carry out daily living tasks.
Time Frame: baseline, 12 months
Population: In the placebo group there were 2 discontinuations (1 moved, 1 death). In the fish oil group there were 2 discontinuations (1 discontinue, 1 death). In the fish oil and lipoic acid group there was 1 discontinuation (due to meds). These discontinuations did not complete the study.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Three 1-gram placebo-fish oil capsule per day and 1 placebo-lipoic acid (LA) capsule per day (600 mg). Placebo fish oil capsules consisted of soybean oil flavored with lemon flavor and 5% fish oil to match fish oil concentrate. LA placebo contained no LA and the following excipients: lactose, hypromellose, silicon dioxide, microcrystalline cellulose, polyethylene glycol, povidone, corn starch, talc, and magnesium stearate.
  Placebo: Soybean oil 3 grams a day and placebo lipoic acid 600 milligrams a day taken for 12 months.
- Fish Oil: Three 1-gram fish oil concentrate capsules in triglyceride form per day (675 mg DHA and 975 mg EPA) and 1 placebo-lipoic acid (LA) capsule (600 mg) per day. LA placebo contained no LA and the following excipients: lactose, hypromellose, silicon dioxide, microcrystalline cellulose, polyethylene glycol, povidone, corn starch, talc, and magnesium stearate.
  Fish Oil: Fish oil concentrate (daily dose 3 grams containing 675 milligrams docosahexanoic acid and 975 milligrams eicosapentanoic acid) taken for 12 months.
- Fish Oil and Lipoic Acid: Three 1-gram fish oil concentrate capsules in triglyceride form per day (675 mg DHA and 975 mg EPA) and 1 lipoic acid (LA) capsule in the racemic form per day (600 mg).
  Fish Oil and Lipoic acid: Fish oil concentrate(daily dose 3 grams containing 675 milligrams docosahexanoic acid and 975 milligrams eicosapentanoic acid) plus lipoic acid (daily dose 600 milligrams)taken for 12 months
Arm/Group | Placebo | Fish Oil | Fish Oil and Lipoic Acid
Number analyzed (Participants) | 11 | 11 | 12
units on a scale | 4.2 (0.9) | 0.7 (1.0) | 0.9 (1.1)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Monthly subject report assessment; prothrombin time and comprehensive metabolic panel at baseline, 6 months, 12 months.
Groups:
- Placebo: Three 1-gram placebo-fish oil capsule per day and 1 placebo-lipoic acid (LA) capsule per day (600 mg). Placebo fish oil capsules consisted of soybean oil flavored with lemon flavor and 5% fish oil to match fish oil concentrate. LA placebo contained no LA and the following excipients: lactose, hypromellose, silicon dioxide, microcrystalline cellulose, polyethylene glycol, povidone, corn starch, talc, and magnesium stearate
- Fish Oil: Three 1-gram fish oil concentrate capsules in triglyceride form per day (675 mg DHA and 975 mg EPA) and 1 placebo-lipoic acid (LA) capsule (600 mg) per day. LA placebo contained no LA and the following excipients: lactose, hypromellose, silicon dioxide, microcrystalline cellulose, polyethylene glycol, povidone, corn starch, talc, and magnesium stearate.
- Fish Oil Plus Lipoic Acid: Three 1-gram fish oil concentrate capsules in triglyceride form per day (675 mg DHA and 975 mg EPA) and 1 lipoic acid (LA) capsule in the racemic form per day (600 mg).
Arm/Group | Placebo | Fish Oil | Fish Oil Plus Lipoic Acid
Serious Adverse Events (participants affected / at risk) | 1/13 | 1/13 | 0/13
Other Adverse Events (participants affected / at risk) | 9/13 | 5/13 | 7/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | Fish Oil (N=13) | Fish Oil Plus Lipoic Acid (N=13)
Heart Failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — death from heart failure subject in fish oil group
Urinary Tract Infection (UTI) (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) — Death resulting from UTI complications in placebo group.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | Fish Oil (N=13) | Fish Oil Plus Lipoic Acid (N=13)
Dizziness (Endocrine disorders) | 1 (1) | 2 (2) | 2 (2)
Falls (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
cold (General disorders) | 3 (3) | 2 (2) | 2 (2)
loose stools (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No